CLINICAL TRIAL: NCT01476995
Title: Prognostic Indicators as Provided by the EPIC ClearView
Acronym: GBMC
Status: Completed | Type: Observational
Sponsor: Epic Research & Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GBMC Triage Study
Record Dates: First submitted 2011-10-03; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Coronary Artery Disease; Congestive Heart Failure; Valvular Heart Disease; Atrial Fibrillation; Hypertension; Pyelonephritis; Acute Renal Failure; Renal Failure; Viral Hepatitis; Alcoholic Hepatitis; Steatohepatitis; Cirrhosis; Asthma; COPD; Bronchitis; Emphysema; Pneumonia; Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Diverticulitis; Peptic Ulcer Disease; Irritable Bowel Syndrome; Cholecystitis; Pancreatitis; Malabsorption Disorders; Celiac Sprue; Diabetes
Keywords: Cardiovascular system; gastrointestinal system; kidneys; liver; lungs
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Heart Valve Diseases; Atrial Fibrillation; Hypertension; Pyelonephritis; Acute Kidney Injury; Renal Insufficiency; Hepatitis, Alcoholic; Fatty Liver; Fibrosis; Asthma; Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema; Pneumonia; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Diverticulitis; Peptic Ulcer; Irritable Bowel Syndrome; Cholecystitis; Pancreatitis; Celiac Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Men and women ages 18-85 lacking any medical diagnosis (as defined in the protocol) of one or more of the following systems/organs: cardiovascular system; gastrointestinal system; kidneys; liver; lungs.
- Five Diagnosis Group: Men and women ages 18-85 with at least one active medical diagnosis (as defined in the protocol) of one or more of the following systems/organs: cardiovascular system; gastrointestinal system; kidneys; liver; lungs.

SUMMARY:
The objective of this study is to determine whether the finger tip images captured by the EPIC ClearView device, when analyzed via the ClearView software, produce a Response Scale that characterizes trends consistent with known diagnoses identified by medical doctors. Specifically, the investigators hypothesize that the organ system involving any of a series of known active diagnoses will be identified in the EPIC ClearView Response Scale report with the intention of providing potential triage capabilities.

ELIGIBILITY:
Inclusion Criteria:

Five Diagnosis Group:

1. Sex: Male or Female
2. Age range: 18 to 85
3. Qualifying medical diagnoses (5 diagnosis groups)

   - For potential subjects presenting with one of the five qualifying diagnoses, the patient presents with confirmed active medical diagnoses affecting the following systems or organs:
   * Cardiovascular system: coronary artery disease, left sided congestive heart failure with EF <50%, valvular heart disease, atrial fibrillation, and hypertension
   * Kidney: pyelonephritis, acute renal failure, or chronic renal failure stages II-V
   * Liver: viral hepatitis, alcoholic hepatitis, steatohepatitis, or cirrhosis
   * Pulmonary system: asthma, COPD, bronchitis, emphysema, or pneumonia
   * Gastrointestinal/Endocrine: inflammatory bowel disease (including Crohn's disease, ulcerative colitis, or diverticulitis), peptic ulcer disease, IBS, cholecystitis, pancreatitis, or malabsorption disorders (including Celiac Sprue); diabetes (Type 1 and Type 2)
4. The patient or legal representative is able to understand and provide signed consent for the procedure.
5. Every effort will be given to balance subjects by gender, age, and race. At least 60 subjects from each of the 5 diagnostic groups and the 1 control group will be recruited.

Control Group:

1. Sex: Male or Female
2. Age range: 18 to 85
3. Freedom from qualifying medical diagnoses (control group)

   - For potential subjects for the control group, the subject is free from active medical diagnoses affecting the following systems or organs:
   * Cardiovascular system: coronary artery disease, left sided congestive heart failure with EF <50%, valvular heart disease, atrial fibrillation, and hypertension
   * Kidney: pyelonephritis, acute renal failure, or chronic renal failure stages II-V
   * Liver: viral hepatitis, alcoholic hepatitis, steatohepatitis, or cirrhosis
   * Pulmonary system: asthma, COPD, bronchitis, emphysema, or pneumonia
   * Gastrointestinal/Endocrine: inflammatory bowel disease (including Crohn's disease, ulcerative colitis, or diverticulitis), peptic ulcer disease, IBS, cholecystitis, pancreatitis, or malabsorption disorders (including Celiac Sprue); diabetes (type 1 and type 2)
4. The patient or legal representative is able to understand and provide signed consent for the procedure.
5. Every effort will be given to balance subjects by gender, age, and race. At least 60 subjects from each of the 5 diagnostic groups and the 1 control group will be recruited.

Exclusion Criteria:

* Patients < 18 years in age or > 85 years in age.
* Inability or unwillingness to provide informed consent.
* Patients with pacemakers or another electrical device implanted somewhere in their body.
* Pregnant women.
* Patients currently undergoing therapy for cancer of any kind.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women ages 18-85 who are inpatients, outpatients, friends/family/staff (controls only) of Greater Baltimore Medical Center in Baltimore, Maryland. Participants cannot have an implantable electrical device (such as a pacemaker) on their body, cannot be pregnant, and cannot be undergoing cancer therapy of any kind.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Agreement of ClearView Scan versus Active Diagnosis | At time of ClearView Scan (Single study visit only, with no follow-up. The study endpoint will be reported for day 0, the day of the study visit).
  Statistical agreement will be assessed between the 0-25 ClearView Response Scale and the physician's diagnoses recorded within the medical record, on a per-subject basis.

SECONDARY OUTCOMES:
Sensitivity and Specificity of ClearView Scan versus Active Diagnosis | Single study visit only, with no follow-up. The study endpoint will be reported for day 0, the day of the study visit.
  Sensitivity and Specificity of the ClearView Scan relative to an active diagnosis, as the proportion of subjects with correctly captured findings amongst those with an active diagnosis and the proportion of subjects without a ClearView finding amongst those without an active diagnosis, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Clair A Francomano, MD, Principal Investigator — Greater Baltimore Medical Center
Locations (1):
- Greater Baltimore Medical Cente, Baltimore, Maryland, United States